CLINICAL TRIAL: NCT01837004
Title: Cognitive Regulation Training and Exercise (CORTEX) Trial
Brief Title: Cognitive Regulation Training and Exercise
Acronym: CORTEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R21HL11341001A1
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-03

CONDITIONS: Patient Compliance
Keywords: adherence; cognition; exercise; aging
MeSH Terms: conditions — Patient Compliance; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- CORTEX (Experimental): The CORTEX group will attend 10, 2-hour sessions for a period of four weeks prior to the initial exercise program start. One hour will be devoted to computerized training (stationary dual-task & cognitive control training, self-priming, certainty training) whereas the other hour will be devoted to exergaming involving non-stationary, dual-task training.
  Interventions: Behavioral: CORTEX

INTERVENTIONS:
Behavioral: CORTEX — 2-hour sessions for a period of four weeks prior to the initial exercise program start. One hour will be devoted to computerized training (stationary dual-task & cognitive control training, self-priming, certainty training) whereas the other hour will be devoted to exergaming involving non-stationary, dual-task training.

SUMMARY:
The purpose of this study is to compare CORTEX (Cognitive Regulation Training and Exercise), a multi-faceted, general and exercise-specific cognitive training program plus a 4-month exercise program, to an attention-control condition involving health and wellness informational lectures plus videos. The proposed exercise program will involve both aerobic and resistive exercises. The investigators hypothesize that pre-intervention cognitive training will enhance self-regulation and self-efficacy and in turn, increase exercise adherence. The investigators also expect more positive improvements in cognitive and psychosocial function among participants in the CORTEX condition as compared to the Control condition immediately following the cognitive booster training, and across time.

DETAILED DESCRIPTION:
Primary Aim 1: To determine the efficacy of pre-intervention cognitive training for improving exercise adherence and engagement. We hypothesize that class participation rates, physical activity counts, and self-reported exercise participation levels will be higher at 4 months for participants in the CORTEX condition relative to the Control condition. We also predict that pre-intervention training will demonstrate high feasibility/acceptability, as indicated by a thorough process evaluation.

Primary Aim 2: To determine if integrated general and exercise-specific cognitive training improves facets of executive function and exercise-related efficacy judgments. We hypothesize that participants in the CORTEX condition will show faster reaction times and greater accuracy for trained and untrained-domain-relevant tasks, including dual task performance, reasoning, and thought-stopping at post-booster testing and 4-month follow-up. Furthermore, we hypothesize that CORTEX participants will show significantly higher levels of exercise efficacy judgments, and exhibit greater automaticity (faster reaction times) in making those judgments, at post-booster testing, 1 month and 4-month follow-up.

Secondary Aim 1: We will use longitudinal mediation analyses to examine mechanisms of change brought about by the cognitive training effects on exercise adherence and engagement. We hypothesize that changes in efficacy and use of self-regulatory strategies will mediate cognitive training effects on exercise adherence over 4-months.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* between 45-64 years old at time of study
* physically inactive for the past 3 months
* have reliable access to internet
* do NOT own or play exergames (Xbox Kinect, Playstation Move, or Nintendo Wii) regularly
* do NOT engage in "brain-training" regularly
* are NOT enrolled in another exercise program or cognitive training study
* willing to be randomized
* able to participant in the full length of the 5-month study with no more than 2 consecutive weeks of vacation

Exclusion Criteria:

* <45 or >64 years of age at time of study
* physically active (i.e., planned 30-min walking or exercise >2 days/wk)
* do not have reliable access to internet
* own and/or play exergames regularly (e.g., 1 day/wk)
* engage in "brain-training" regularly (e.g., Sudoku or computer game-play 1 day/wk)
* enrolled in another exercise program or cognitive training study
* cognitive impairment as defined by TICS score <21
* depression as defined by Geriatric Depression Scale score >5

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
exercise adherence | 4 months (from exercise intervention baseline to 4-month post-test)
  * number of weekly classes attended (out of 16 total)
  * frequency of electronically-recorded visits to the fitness facility
exercise program engagement | 4 month period (exercise intervention start to end)
  * self-reported physical activity
  * activity counts assessed via accelerometer
  * weekly exercise logs
  * website usage & percentage of online educational modules completed

SECONDARY OUTCOMES:
automaticity of exercise-related efficacy judgments | 5-month period
  -reaction times and interference associated with a novel self-efficacy judgment task; collected at baseline, m1, and m5
exercise-related self-efficacy | 5-month period
  -self-reported confidence in one's ability to adhere to different aspects of the exercise program; collected at baseline, m1, m2, and m5
executive functioning | 5-month period
  -trained and untrained domains of executive functioning (e.g., dual-task ability, inhibitory control, reasoning) and memory assessed via computer-based and pencil-paper tasks; collected at baseline, 1m, and 5m

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Mullen, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois, Urbana, Illinois, United States